## Postpregnancy Family Planning Choices in Public and Private Sectors in Kenya and Indonesia (PPFP Choices)

Statistical Analysis Plan

Jhpiego

Unique Protocol ID: IRB00007462

October 31, 2017

Uploaded to Clinicaltrials.gov on November 2, 2017

## **Data Analysis Plan**

## Postpregnancy Family Planning Choices in Public and Private Sectors in Kenya and Indonesia (PPFP Choices)

The data analysis plan describes how data collected through different methods will be analyzed after cleaning in order to answer the research questions. Overall, triangulation of findings from quantitative and qualitative data analysis will be done to ensure that the findings provide deeper insights into the study objectives.

- A. <u>Client Interviews Data Analysis</u>: Descriptive statistics will be done, computing means and standard deviations for continuous variables and percentages for categorical variables: Proportion of pregnant/postpartum women who choose a FP method during antenatal care (ANC) or early labor, and, of those, what proportion received the FP method in the immediate postpregnancy period (prior to discharge). In addition, logistic **bivariare and multivariavle regression** will be used to explore differences in acceptance of PPFP between the intervention and control facilities, A p-value of <0.05 will be considered statistically significant in bivariate analysis for variables to be selected for inclusion in **multilevel analysis** model to determine the factors affecting intention to use and receipt of PPFP.
- B. Key Informant interviews, Focus Group Discussions and In-Depth Interviews: Data will all be analyzed using Grounded Theory methods. Initial KII, FGD and IDI responses will be translated, transcribed, coded, and analyzed using software to facilitate data management. Quality of translation will be checked for each (KIIs, FGDs and IDIs) through back translation of a randomly-selected subset of 6 interviews. Using Atlas.TI analytical software, coding will be used to conceptually name the data and reduce it to manageable units of information that cover broad and general categories. A priori codes will be developed based on the concepts of interest in this research (perception of risk, benefits and beliefs, etc.) and the study aims. As additional KIIs, FGDs and IDIs are conducted, these a priori codes will be complemented by additional codes that reflect themes and concepts that emerge from the data. Codebooks will be developed for the different concepts to facilitate consistency in the coding process. The coded data will be organized into a hierarchy of themes which are then meaningfully linked to each other to show patterns, relationships and explanations. In conjunction with the coding process, memos will be used to develop conceptual categories and themes and to track emerging insights and interpretations].
- C. <u>Family Planning Facility Registers:</u> Using FP Facility Register data, the study team will assess trends in service delivery at participating facilities including the total number of ANC clients, the total number of Labor and Delivery clients, total number of postabortion clients, the total number of postpartum family planning acceptors broken into the type of family planning method accepted. Additionally, the study and project teams will monitor facility records for reports of adverse events related to PPFP acceptance.
- D. <u>Supportive Supervision Records</u>: Supportive Supervision Records will primarily be used to measure changes in service provision quality according to data collected during the Supportive Supervision. Overall changes in the number/percent of standards met will be calculated through difference in difference analysis. Facility aggregate provider performance information may also be calculated into assessment of facility readiness and overall facility quality.

E. <u>Facility Audits Data Analysis:</u> Mapping of facilities will be visually analyzed to provide further understanding of structural issues that may influence perceptions and key behaviors. Aggregated country and district/county data from the baseline audits will be used to inform final program intervention design where possible. Additionally, select data from the client interviews will be combined with key facility level indicators for a **multilevel analysis** of the factors affecting intention to use and receipt of immediate post-pregnancy family planning methods, and to assess the overall success of the program.